CLINICAL TRIAL: NCT05314179
Title: Ubuntu - I Am Because We Are, Caring for Black Patients With Advanced Stage Cancer
Brief Title: Ubuntu - I Am Because We Are
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Margaret Quinn Rosenzweig, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HCC 21-265
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Cancer
Keywords: doula
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Pre and post intervention pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doula-Patient engagement (Experimental): Four hours/week of Ubuntu ambassador/Doula and Patient engagement. The nature and type of visits will be determined by the patient and doula.
  The doula will formulate weekly reports for each assigned patient. Weekly progress reporting - Weeks 2- 24.
  Interventions: Behavioral: Doula - Patient engagement

INTERVENTIONS:
Behavioral: Doula - Patient engagement — Ubuntu ambassador/Doula and Patient will decide on details of engagement. The components to be included will be: 1) emotional support, 2) practical assistance, 3) family support, and/or 4) legacy building projects as per study protocols.
  The nature and type of visits will be determined by the patient and doula.

SUMMARY:
The program will provide Advocacy and Support for Black patients with advanced-stage cancer in the Pittsburgh area. The goals are to: 1) provide a community-based, trained companion to journey alongside the patient with advanced cancer, 2) to help the individual explore meaning and create legacy, 3); offer support and navigation for practical needs of illness (e.g., financial assistance for food and housing, accessing and affording medications, transportation); and 4) to provide support and connection for the bereaved family/friends, including facilitating community connections for routine health screenings and access to mental health services, as needed.

DETAILED DESCRIPTION:
Across almost all types of cancer, Black patients experience shorter survival and disproportionate burdens of isolation, pain, financial toxicity, and symptom distress at the end of life. The importance of palliative care in providing patient-centered treatment plans that alleviate symptom burden and provide goal-concordant care is well-established; however, Black patients have been historically reluctant to utilize traditional palliative care and hospice services despite efforts on the part of the largely white palliative care community to increase their utilization. This proposed program provides a non-medically focused program to assist Black patients living with advanced cancer. Black individuals are less likely to discuss their end-of-life (EOL) plans before death (1), engage in advanced care planning, use hospice (2), and are more likely to undergo intensive treatment in the last months of life (2-4), limiting the ability of the patient and family to receive an end of life support and create a legacy. Low-income black individuals have additional practical needs for food, housing, transportation, and medication assistance exacerbated by the advanced illness often overwhelming the traditional assistance capabilities of the medical model. There is a growing need for innovation to meet the EOL care needs of Black populations and communities requiring more culturally tailored support than traditionally available from the cancer care delivery system.

The goal is to provide

1. a community-based, peer, trained, paid companion to journey alongside the patient with advanced cancer, providing support, advocacy, and acknowledgment of the fear and trauma of living with a progressive, life-ending illness,
2. to help the individual recognize their unique legacy,
3. to assist surviving family members with mental and physical health promotion. The navigators/social workers or community advocates will identify individuals/patients who are eligible for the study. If the advocate is able to be at the clinic site at the time of the appointment, they will meet with the patient to say hello if the patient agrees. They will speak to the patient/family about the program. Patients will be asked if the ambassadors can call and make the connection.

ELIGIBILITY:
Inclusion Criteria:

1. have stage IV cancer
2. identify as Black or African American 3. Participants must reside in or around Pittsburgh, Pennsylvania area

Exclusion Criteria:

1. Do not live in the Pittsburgh region

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2022-03-13 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Change in Integrated Palliative care Outcome Scale (IPOS) | Baseline, 3 months and 6 months
  IPOS (Integrated Palliative care Outcome Scale) is a measure of symptoms and concerns which matter to a patient and helps us provide the best care. IPOS forms to identify how we can best support the individual. There are 10 questions scored on a scale of 1-4, which assess a patient's symptoms and needs with regards to physical, social, psychological and spiritual. Higher scores indicate greater patient need for supportive care.
Acceptability and feasibility of the Doula Program | Up to 6 months
  Acceptability and feasibility of doula program will be assessed by the Evaluation of the UPP Program questionnaire, which is comprised of 7 questions that will be used to rate participant satisfaction with the Doula Program that employ a scale of 1 (not at all) to 10 (to a great degree). Higher overall scores indicate greater satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Quinn Rosenzweig, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No